CLINICAL TRIAL: NCT01571466
Title: A Double-blind Phase I Study to Evaluate the Safety of the HIV-1 Vaccine MVA-B in Chronic HIV-1 Infected Patients Successfully Treated With HAART
Brief Title: A Study to Evaluate the Safety of the HIV-1 Vaccine MVA-B in Chronic HIV-1 Infected Patients Successfully Treated With HAART
Acronym: 2009-016578-34
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Felipe Garcia, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RisVac 03
Record Dates: First submitted 2011-11-09; First posted 2012-04-05 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine group (Experimental): Modified Pox virus, strain MVA clade -B (expressing HIV-1 Bx08gp120 and IIIB gagpolnef) (MVA HIV-B)
  Interventions: Drug: Vaccination
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaccination — * Modified Pox virus, strain MVA clade -B (expressing HIV-1 Bx08gp120 and IIIB gagpolnef)
    -~ 1 x 10e8 pfu/ml
  * 3 immunisations at week 0, 4 and 16
  Arms: Vaccine group
Drug: Placebo — 3 immunisations at week 0, 4 and 16
  Arms: Placebo

SUMMARY:
30 treated chronic HIV-1 infected patients with CD4+ cell counts above 450 cells/ mm3 will be randomized 1:2 to receive placebo (n=10) or vaccine (n=20) at week 0, 4 and 16 and will be observed at the Investigation Unit of the study site for one hour following vaccination. At week 24 they will stop their HAART until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age;
* Voluntarily signed informed consent;
* Patient is male, or female with negative pregnancy test prior to enrolment;
* Patient has a proven HIV-1 infection (with positive antibodies against HIV-1 and a detectable plasma HIV-1 RNA);
* Patient must be on stable treatment with HAART for at least 6 months (HAART is defined as an antiretroviral regimen consisting of at least three registered antiretroviral agents*);
* Mean of all measured CD4+ cell counts during the 6 months prior to the start of HAART must be above or equal to 200 cells/ mm3
* Current CD4+ cell count must be at least 450 cells/ mm3;
* HIV-RNA must be below 50 copies/ mL for the last 6 months prior to inclusion, during at least two measurements (occasional so called 'blips' up to 50 copies/mL are permitted);
* Patient is one of the following: not sexually active, or a heterosexually active female, agreeing to use condoms with her partner from 14 days prior to the first vaccination until 4 months after the last, even though using another method of contraception, and willing to undergo pregnancy tests during screening and prior to each vaccination, or a male, agreeing to use condoms with his partner from the day of the first vaccination until 4 months after the last vaccination.

Exclusion Criteria:

* Treatment with a non-HAART regimen of antiretroviral agents prior to the start of HAART;
* History of a CDC class C event (see Appendix);
* Interruption of HAART during the course of the study which is expected at the time of inclusion;
* History of exposure <20 years ago to any poxvirus based vaccine;
* Patient is female and has a positive pregnancy test or the wish of pregnancy:
* Active opportunistic infection, or any active infection or malignancy within 30 days prior to screening visit;
* Therapy with immunomodulatory agents, including cytokines (e.g. IL2) and gamma globulin, or cytostatic chemotherapy within 90 days prior to screening visit;
* History of allergy to any vaccine component;
* Use of anti-coagulant medication;
* Use of any investigational drug during the 90 days prior to study entry;
* Previous failure to antiretroviral and/or mutations conferring genotypic resistance to antiretroviral therapy
* Any other condition which, in the opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
primary safety parameters | week 8
  Grade 3 or above local adverse event (pain, cutaneous reactions including induration) Grade 3 or above systemic adverse event (temperature, chills, headache, nausea, vomiting, malaise, and myalgia) Grade 3 or above other clinical or laboratory adverse event confirmed at examination or on repeat testing respectively Any event attributable to vaccine leading to discontinuation of the immunisation regimen
Primary immunogenicity parameters | After each inmunisation and at weeks 6-8 and 18-20
  Cellular responses - CD8/CD4+ T cell responses (ELISPOT)

SECONDARY OUTCOMES:
All grade 1 and 2 adverse events | week 8
Viral load rebound | week 48
  After HAART interruption compared between both arms and with baseline viral load before any medication in each arm
Antibody responses | 48 weeks
  * binding titration to the construct MVAB
  * binding titration to and neutralisation of vaccinia
Cellular responses | Week 6 and 18
  Intracellular cytokine analysis

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid

REFERENCES:
- [Derived] Gomez CE, Perdiguero B, Garcia-Arriaza J, Cepeda V, Sanchez-Sorzano CO, Mothe B, Jimenez JL, Munoz-Fernandez MA, Gatell JM, Lopez Bernaldo de Quiros JC, Brander C, Garcia F, Esteban M. A Phase I Randomized Therapeutic MVA-B Vaccination Improves the Magnitude and Quality of the T Cell Immune Responses in HIV-1-Infected Subjects on HAART. PLoS One. 2015 Nov 6;10(11):e0141456. doi: 10.1371/journal.pone.0141456. eCollection 2015. PMID 26544853
- [Derived] Mothe B, Climent N, Plana M, Rosas M, Jimenez JL, Munoz-Fernandez MA, Puertas MC, Carrillo J, Gonzalez N, Leon A, Pich J, Arnaiz JA, Gatell JM, Clotet B, Blanco J, Alcami J, Martinez-Picado J, Alvarez-Fernandez C, Sanchez-Palomino S, Guardo AC, Pena J, Benito JM, Rallon N, Gomez CE, Perdiguero B, Garcia-Arriaza J, Esteban M, Lopez Bernaldo de Quiros JC, Brander C, Garcia F; RISVAC-03 Study Group. Safety and immunogenicity of a modified vaccinia Ankara-based HIV-1 vaccine (MVA-B) in HIV-1-infected patients alone or in combination with a drug to reactivate latent HIV-1. J Antimicrob Chemother. 2015;70(6):1833-42. doi: 10.1093/jac/dkv046. Epub 2015 Feb 26. PMID 25724985